CLINICAL TRIAL: NCT05447208
Title: A Randomized Control Trial to Investigate the Effect of Growth Hormone on the Euploid Rate of Blastocyst in Patients With Advanced Maternal Age
Brief Title: Effect of GH on the Blastocyst Euploid Rate in AMA Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022JIAI-10
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Preimplantation Genetic Testing; Growth Hormone; Age, Parental
MeSH Terms: interventions — Growth Hormone; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The embryologists, genetic scientists, and the independent statistician will be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): GH is supplemented during ovarian stimulation
  Interventions: Drug: Growth Hormone; Drug: GnRH antagonist
- Control group (Active Comparator): GH is not supplemented during ovarian stimulation.
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: Growth Hormone — Growth hormone is supplemented before and during the ovarian stimulation till the day of oocyte retrieval
  Arms: Treatment group
Drug: GnRH antagonist — GnRH antagonist (Cetrorelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger

SUMMARY:
This randomized trial aims to compare the euploid rate of blastocysts in AMA patients undergoing PGT-A (preimplantation genetic testing for aneuploidy) with or without growth hormone supplement.

Infertile patients ≥38 years old will be recruited for study after informed consent if they fulfill the inclusion criteria and do not have the exclusion criteria. Eligible women will be randomised into one of the two groups:

Treatment group: Women will receive growth hormone (GH) supplement before and during antagonist protocol for ovarian stimulation.

Control group: Women will receive antagonist protocol for ovarian stimulation. The primary outcome is the euploidy rate of blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥38; intended to undergo PGT-A
* BMI in the normal range (18.50-24.0kg/m2)
* Normal semen analysis for the male partner

Exclusion Criteria:

* Endometriosis grade 3 or higher, untreat hydrosalpinx
* Women with a uterine cavity abnormality, such as a uterine congenital malformation (uterus uni-cornate, bicornate, or duplex); untreated uterine septum, adenomyosis, submucous myoma, or endo-metrial polyp(s)
* Women who are indicated and planned to undergo PGT-SR (Preimplantation genetic testing for structural rearrangement) or PGT-M (Preimplantation genetic testing for monogenic disorder), for example, parental abnormal karyo-type or diagnosed with monogenic disease
* History of endocrine disorder, autoimmune diseases or diagnosed thrombophilia
* History of GH supplementation in the previous IVF treatment or taking other supplementary drugs used during stimulation; patients with absolute or relative contraindications to GH treatment, including active malignancy or history of cancer, diabetic retinopathy, diabetes mellitus, and chronic kidney disease.

Min Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
euploidy rate | 1 month after oocyte retrieval
  euploidy rate of blastocysts

SECONDARY OUTCOMES:
live birth rate | 1 year after embryo transfer
  deliveries ≥22 weeks gestation with heartbeat and breath of the first frozen embryo transfer
cumulative live birth rate | 1 year after embryo transfer
  cumulative live birth within 6 months of randomization
ongoing pregnancy | 12 weeks' gestation
  a viable pregnancy beyond 12 weeks' gestation of the first frozen embryo transfer
clinical pregnancy rate | 6 weeks after embryo transfer
  the presence of intrauterine gestational sac by transvaginal ultrasound at 6 gestational weeks of the first frozen embryo transfer
number of euploid blastocysts in an OS cycle | 1 month after oocyte retrieval
  the number of blastocysts acquired in an ovarian stimulation cycle that are identified as euploid by PGT-A
the probability of obtaining euploid blastocysts in an OS cycle | 1 month after oocyte retrieval
  If the ovarian stimulation cycle produces euploid blastocysts, the result is 1; if not, it's 0. Mean values will be calculated for the two groups.
KIDScore of euploid embryos | 6 days after oocyte retrieval
  an AI-driven embryo score generated through the EmbryoViewer software relying on kinetic parameters and associated with embryo implantation potential

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PhD, Principal Investigator — Shanghai JiAi Genetics & IVF Institute, China
Locations (1):
- Shanghai JIAI Genetics and IVF Institute, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available when beginning 3 months and ending 5 years following article publication
Access Criteria: To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with. Proposals should be sent to 08301010255@fudan.edu.cn.

REFERENCES:
- [Background] Demko ZP, Simon AL, McCoy RC, Petrov DA, Rabinowitz M. Effects of maternal age on euploidy rates in a large cohort of embryos analyzed with 24-chromosome single-nucleotide polymorphism-based preimplantation genetic screening. Fertil Steril. 2016 May;105(5):1307-1313. doi: 10.1016/j.fertnstert.2016.01.025. Epub 2016 Feb 8. PMID 26868992
- [Background] Weall BM, Al-Samerria S, Conceicao J, Yovich JL, Almahbobi G. A direct action for GH in improvement of oocyte quality in poor-responder patients. Reproduction. 2015 Feb;149(2):147-54. doi: 10.1530/REP-14-0494. Epub 2014 Nov 5. PMID 25376626
- [Background] Gong Y, Luo S, Fan P, Jin S, Zhu H, Deng T, Quan Y, Huang W. Growth hormone alleviates oxidative stress and improves oocyte quality in Chinese women with polycystic ovary syndrome: a randomized controlled trial. Sci Rep. 2020 Oct 30;10(1):18769. doi: 10.1038/s41598-020-75107-4. PMID 33127971
- [Background] Liu C, Li S, Li Y, Tian J, Sun X, Song T, Yan G, Ding L, Sun H. Growth hormone ameliorates the age-associated depletion of ovarian reserve and decline of oocyte quality via inhibiting the activation of Fos and Jun signaling. Aging (Albany NY). 2021 Feb 17;13(5):6765-6781. doi: 10.18632/aging.202534. Epub 2021 Feb 17. PMID 33621201
- [Background] Skillern A, Leonard W, Pike J, Mak W. Growth hormone supplementation during ovarian stimulation improves oocyte and embryo outcomes in IVF/PGT-A cycles of women who are not poor responders. J Assist Reprod Genet. 2021 May;38(5):1055-1060. doi: 10.1007/s10815-021-02088-2. Epub 2021 Feb 3. PMID 33534048
- [Background] Regan SLP, Knight PG, Yovich JL, Arfuso F, Dharmarajan A. Growth hormone during in vitro fertilization in older women modulates the density of receptors in granulosa cells, with improved pregnancy outcomes. Fertil Steril. 2018 Dec;110(7):1298-1310. doi: 10.1016/j.fertnstert.2018.08.018. PMID 30503129